CLINICAL TRIAL: NCT00629226
Title: Phase I Study of Bortezomib and Cetuximab Without or With Cisplatin in Combination With Radiation Therapy for Advanced Head and Neck Cancer
Brief Title: Bortezomib, Cetuximab, and Radiation Therapy With or Without Cisplatin in Treating Patients With Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 080071, CDR0000588196; NCI-08-C-0071; CCR 7205; NCI-7893
Record Dates: First submitted 2008-03-01; First posted 2008-03-05 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Bortezomib; Cisplatin; Radiotherapy, Intensity-Modulated

ARMS (2):
- Group I (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, and 50. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, 11, 22, 25, 29, 32, 43, 46, 50, and 53. Beginning on day 8 or 9, patients undergo standard intensity-modulated radiotherapy (IMRT) once daily, 5 days a week, for up to 8 weeks.
  Interventions: Biological: cetuximab; Drug: bortezomib; Radiation: intensity-modulated radiation therapy
- Group II (Experimental): Patients receive cetuximab, bortezomib (beginning at one dose level below the MTD determined in group I), and IMRT as in group I. Patients also receive cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, and 57.
  Interventions: Biological: cetuximab; Drug: bortezomib; Drug: cisplatin; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: cetuximab — Given IV
Drug: bortezomib — Given IV
Drug: cisplatin — Given IV
  Arms: Group II
Radiation: intensity-modulated radiation therapy — Once daily, 5 days a week, for up to 8 weeks

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high energy x- rays to kill tumor cells. Bortezomib and cetuximab may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with cetuximab, radiation therapy, and cisplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with cetuximab and radiation therapy with or without cisplatin in treating patients with stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility and toxicity of bortezomib, cetuximab, and radiotherapy with or without cisplatin in patients with stage IV squamous cell carcinoma of the head and neck.
* To identify the maximum tolerated dose of bortezomib for further clinical phase II development.

Secondary

* To evaluate the objective response rate, progression-free survival, and overall survival of patients treated with these regimens.
* To determine the effects of bortezomib and cetuximab with or without cisplatin on inhibiting activation of the NF-kB, EGFR, MAPK, and STAT3 signal pathways, expression of pro-survival and pro-angiogenesis genes regulated by these pathways, and on proliferation, apoptosis, and angiogenesis.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib. Patients are simultaneously accrued to 1 of 2 treatment groups. Patients are initially accrued to group I until there are a sufficient number of patients to establish the maximum tolerated dose (MTD) of bortezomib. Patients are then accrued to group II.

* Group I: Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, and 50. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, 11, 22, 25, 29, 32, 43, 46, 50, and 53. Beginning on day 8 or 9, patients undergo standard intensity-modulated radiotherapy (IMRT) once daily, 5 days a week, for up to 8 weeks.

Once the MTD of bortezomib is determined, at least 6 and up to 10 additional patients are accrued and treated at the MTD.

* Group II: Patients receive cetuximab, bortezomib (beginning at one dose level below the MTD determined in group I), and IMRT as in group I. Patients also receive cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, and 57.

Once the MTD of bortezomib is determined, 6 additional patients are accrued and treated at the MTD.

Patients undergo blood sample collection periodically for correlative laboratory studies. Samples are analyzed for biomarkers by immunohistochemistry, quantitative reverse transcriptase-polymerase chain reaction, and ELISA.

After completion of study therapy, patients are followed periodically for 2-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck, including variants or undifferentiated/poorly differentiated carcinoma

  * Previously untreated stage IV disease OR residual disease or regionally recurrent disease after prior surgery and/or chemotherapy
* Must be eligible to receive full-dose radiotherapy and be evaluated and accepted for treatment by a Radiation Oncologist
* No clinically measurable distant disease OR has asymptomatic small distant lesions outside the radiation field ≤ 3 cm in individual or aggregate diameter for which palliation of local and regional disease is clearly warranted
* No previously untreated nasopharyngeal cancer (any stage)

  * Recurrent nasopharyngeal carcinoma allowed
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* ANC ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Total bilirubin normal (indirect bilirubin ≤ 3 mg/dL in patients with Gilbert's syndrome)
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate cognitive and neurologic function
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, cetuximab, cisplatin, or other agents used in this study
* No peripheral sensory neuropathy ≥ grade 2
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would preclude study compliance
* HIV-negative

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 3 months since prior cisplatin
* No prior radiotherapy to the head and neck
* No prior systemic EGFR inhibitors
* No prior bortezomib
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent antiretroviral therapy
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and other toxicities as assessed by NCI CTCAE v3.0
Maximum tolerated dose of bortezomib when administered in combination with cetuximab and radiotherapy with and without cisplatin

SECONDARY OUTCOMES:
Objective response rate
Progression-free survival
Overall survival
Pre-to-post-treatment changes in biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Carter Van Waes, MD, PhD, Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania